CLINICAL TRIAL: NCT04325672
Title: Convalescent Plasma to Limit Coronavirus Associated Complications: An Open Label, Phase 2A Study of High-Titer Anti-SARS-CoV-2 Plasma in Hospitalized Patients With COVID-19
Brief Title: Convalescent Plasma to Limit Coronavirus Associated Complications
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: Study stopped due to opening Expanded Access Protocol.
Sponsor: Mayo Clinic (Other)
Responsible Party: Principal Investigator, Michael J. Joyner, M.D., Principal Investigator, Mayo Clinic
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 20-002864
Record Dates: First submitted 2020-03-26; First posted 2020-03-27 (Actual); Last update posted 2020-04-08 (Actual); Status verified 2020-04

CONDITIONS: Coronavirus
Keywords: 2019 novel Coronavirus; SARS-CoV-2; COVID-19
MeSH Terms: conditions — Coronavirus Infections; COVID-19

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Convalescent Plasma Group (Experimental): Subjects will receive 1-2 units (300-600 mL) of plasma with an anti-SARS-CoV-2 titer of >1:64.
  Interventions: Biological: Convalescent Plasma

INTERVENTIONS:
Biological: Convalescent Plasma — Anti-SARS-CoV-2 convalescent plasma obtained from patients identified as having recovered from COVID-19 with neutralizing antibody titers >1:64.

SUMMARY:
Researchers are trying to assess the treatment potential and safety of anti-SARS-CoV-2 convalescent plasma in patients with acute respiratory symptoms with confirmed COVID-19.

DETAILED DESCRIPTION:
High titer human convalescent plasma will be extracted from apheresis donations from twenty recently-sick and currently-recovered COVID-19 patients. An open-label, phase 2A clinical trial will then be conducted to administer convalescent plasma to twenty individuals with confirmed cases of COVID-19 to investigate the novel application of convalescent plasma in the treatment strategy of SARS-CoV-2.

ELIGIBILITY:
Inclusion Criteria:

* Patients must be 18 years of age or older
* Hospitalized with COVID-19 respiratory symptoms and confirmation via COVID-19 SARS-CoV-2 RT-PCR testing. Patient is willing and able to provide written informed consent and comply with all protocol requirements.
* Patient agrees to storage of specimens for future testing.

Exclusion Criteria:

* Female subjects with positive pregnancy test, breastfeeding, or planning to become pregnant/breastfeed during the study period
* Receipt of pooled immunoglobulin in past 30 days
* Contraindication to transfusion or history of prior reactions to transfusion blood products

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2020-04-01 (Estimated); Primary Completion 2022-12-31 (Estimated); Study Completion 2022-12-31 (Estimated)

PRIMARY OUTCOMES:
RNA in SARS-CoV-2 | Days 0, 1, 3, 7, 14, 28, 60 and 90 after transfusion
  Change in RNA levels of SARS-CoV-2 from nasopharyngeal using RT-PCR (reverse transcriptase polymerase chain reaction) across time.
ICU Admissions | 90 days after transfusion
  Total number of subjects to be admitted to the ICU after the anti-SARS-CoV-2 convalescent plasma transfusion.
Hospital Mortality | 90 days after transfusion
  Total number of subject deaths.
Hospital Length of Stay (LOS) | 90 days after transfusion
  The total number of days subjects were admitted to the hospital.

SECONDARY OUTCOMES:
Type of respiratory support | 90 days after transfusion or until hospital discharge (whichever comes first)
  The type of supplemental oxygen support (e.g. nasal cannula, high flow nasal cannula, noninvasive ventilation, intubation and invasive mechanical ventilation, rescue ventilation) of the anti-SARS-CoV-2 convalescent plasma group across time.
Duration of respiratory support | 90 days after transfusion or until hospital discharge (whichever comes first)
  The total number of days subjects required respiratory support.

CONTACTS AND LOCATIONS:
Overall Officials: Michael Joyner, MD, Principal Investigator — Mayo Clinic

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Mayo Clinic Clinical Trials — https://www.mayo.edu/research/clinical-trials